CLINICAL TRIAL: NCT06831097
Title: Early Childhood Obesity Among Rural Residents of West Texas
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University Health Sciences Center (Other)
Collaborators: University of Nevada, Las Vegas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 25-0166
Record Dates: First submitted 2025-02-03; First posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Obesity
Keywords: Obesity; Children; Obesity prevention in children
MeSH Terms: conditions — Obesity | interventions — Food; Health; Gardens

STUDY DESIGN:
Intervention Model Description: In this 5-year project, a longitudinal CBPR research design and a mixed method approach will be employed. We will use a group randomized trial (GRT) with two arms (an intervention arm and a wait-list control arm) to test the effectiveness of the Para Salud interventions compared to usual care received from the Head Start (HS) programs, because children are nested in class at the HS centers and the Pasos Para Salud intervention will be delivered in in classrooms. Data will be collected pre-intervention, at the mid-point intra-intervention, immediately post-intervention, and 6 and 12 months post-intervention. Cohort 1 will consist of the four rural sites from Terry, Hockley, Lamb and Lubbock counties. We will add Cohort 2 consisting of HS students from Hale, Floyd, Crosby, Garza and Lynn counties in project Y3.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- wait-list control (No Intervention): Usual Head Start activities
- Para Salud (Experimental): Arm Description: "Comidas Para Salud" (Food for Health), will focus on assisting young children to learn skills in healthy eating. The Bienestar Preschool Curriculum is home-based and directed to both the primary caregivers as well as the child participants. The "Pasos Para Salud" (Steps for Health), which will use IVG/exergaming to increase children's physical activity level and reduce their sedentary behavior. "Jardines Para Salud" (Gardens for Health), will involve planting gardens in the HS settings and supervised home gardening projects for the preschool participants and their parents/guardians. This will instill the value of gardening and gardening skills in promoting a healthy lifestyle.
  Interventions: Behavioral: "Comidas Para Salud" (Food for Health), "Pasos Para Salud" (Steps for Health), "Jardines Para Salud" (Gardens for Health)

INTERVENTIONS:
Behavioral: "Comidas Para Salud" (Food for Health), "Pasos Para Salud" (Steps for Health), "Jardines Para Salud" (Gardens for Health) — "Comidas Para Salud" (Food for Health), "Pasos Para Salud" (Steps for Health), "Jardines Para Salud" (Gardens for Health)
  Description: Arm Description: "Comidas Para Salud" (Food for Health), will focus on assisting young children to learn skills in healthy eating. The Bienestar Preschool Curriculum is home-based and directed to both the primary caregivers as well as the child participants. The "Pasos Para Salud" (Steps for Health), which will use IVG/exergaming to increase children's physical activity level and reduce their sedentary behavior. "Jardines Para Salud" (Gardens for Health), will involve planting gardens in the HS settings and supervised home gardening projects for the preschool participants and their parents/guardians. This will instill the value of gardening and gardening skills in promoting a healthy lifestyle.
  Arms: Para Salud

SUMMARY:
The Para Salud study is a longitudinal, community-based participatory research (CBPR) initiative aimed at preventing and controlling obesity among preschool children in rural Texas. The study will implement evidence-based interventions targeting nutrition, physical activity, and gardening. The interventions are designed to improve health outcomes, specifically in reducing obesity-related metrics among young Hispanic children, who are at a higher risk of obesity due to social determinants of health.

Primary Objective: To assess the effectiveness of the Para Salud interventions in reducing obesity-related metrics, including BMI percentile, waist-to-height ratio, and percentage body fat, among preschool children aged 3-4 years in the Texas High Plains over a 24-month period.

Secondary Objective: To evaluate the impact of the Para Salud interventions on increasing physical activity levels, improving dietary habits (such as increasing fruit and vegetable intake), and reducing sedentary behavior and sugar-sweetened beverage consumption among the study participants.

DETAILED DESCRIPTION:
The study will enroll 480 children aged 3-4 years from Head Start (HS) programs in the rural areas of Crosby, Floyd, Garza, Hale, Hockley, Lamb, Lubbock, Lynn, and Terry counties, Texas. The population is predominantly Hispanic and of low socioeconomic status, with a significant proportion living in medically underserved areas.

The study is in the implementation and evaluation phase, focusing on interventions aimed at preventing and controlling obesity in a specific high-risk population of preschool-aged children in rural Texas.

Participants will be enrolled from Head Start (HS) programs in nine counties: Crosby, Floyd, Garza, Hale, Hockley, Lamb, Lubbock, Lynn, and Terry. The study will be directed through the School of Nursing (SON) at Texas Tech University Health Sciences Center, specifically through the Larry Combest Community Health and Wellness Center (LCCHWC), a nurse-led federally-qualified health center located in East Lubbock. If needed, the LCCHWC has established facilities for implementing the study interventions, including classrooms for nutrition educational and physical activity programs and spaces for gardening projects, having been a primary site for the USDA-funded research project.

Comidas Para Salud (Food for Health): Nutrition education and home-based interventions to teach healthy eating habits.

Pasos Para Salud (Steps for Health): Physical activity intervention using interactive video gaming to increase daily physical activity and reduce sedentary behavior.

Jardines Para Salud (Gardens for Health): Gardening activities conducted at both school and home to promote physical activity and healthy eating through hands-on experiences in growing fruits and vegetables.

The overall study duration is 5 years, including recruitment, intervention implementation, and follow-up assessments.

Each participant will be involved in the study for 24 months, which includes baseline assessments, 12 months of intervention, and follow-up assessments at 6 and 12 months post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in the participating HS programs,
* Aged 3-4 years,
* Live in a selected county in Texas High Plains (Crosby, Floyd, Garza, Hale, Hockley, Lamb, Lubbock, Lynn, and Terry County)
* Without a diagnosed physical or mental disability according to enrollment records,
* Parental consent
* The inclusion criteria will be verified through children's enrollment records and the demographic information sheet. The parental/guardian participants will be the primary caregiver of each participating child, who lives in the same household of the child.

Exclusion Criteria:

* Health Status: Children with diagnosed physical or mental disabilities according to enrollment records.
* Lack of Consent: Children without parental/guardian consent to participate in the study.

Ages: 3 Years to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 480 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2030-03-30 (Estimated); Study Completion 2030-08-30 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome 1 | Baseline (T0), 6 months (T1.), 12 months (T2), and follow-ups at 6 and 12 months after the intervention starts for the control group
  Height and Weight: These will be measured using a stadiometer and electronic scale (Tanita). The measurements will include Body Mass Index (BMI) percentile adjusted for age and gender, as well as body fat percentage.
Primary Outcome 2 | Baseline (T0), 6 months (T1.), 12 months (T2), and follow-ups at 6 and 12 months after the intervention starts for the control group
  Waist Circumference (WC) and Waist-to-Height Ratio (WHTR): WC will be measured at the top of the right ilium, and WHTR will be calculated.
Primary Outcome 3 | Baseline (T0), 6 months (T1), 12 months (T2), and follow-ups at 6 and 12 months after the intervention starts for the control group.
  A self-administered survey will collect demographic, socioeconomic, and lifestyle data, including TV in the bedroom, screen time, parental support for physical activity, sugar-sweetened beverage intake, fruit and vegetable intake, frequency of family meals, and fast food consumption.
Primary Outcome 4 | Baseline (T0), 6 months (T1), 12 months (T2), and follow-ups at 6 and 12 months after the intervention starts for the control group
  Nutrition Knowledge: This will be assessed using the Nutritional Knowledge Assessment (NKT), which includes questions on energy intake, nutrient content, and food knowledge.
Primary Outcome 5 | Baseline (T0), 6 months (T1), 12 months (T2), and follow-ups at 6 and 12 months after the intervention starts for the control group
  Physical activity levels will be assessed using ActiGraph accelerometers, which will record daily activity counts and categorize them into sedentary, light, moderate, and vigorous levels.

CONTACTS AND LOCATIONS:
Locations (1):
- Texas Tech University Health Sciences Center, Lubbock, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
We will be meeting with the Community Advisory Board before this decision will be made.